CLINICAL TRIAL: NCT02895321
Title: Randomized Clinical Trial to Evaluate the Efficacy of Nano-hydroxyapatite Combined With the Potassium Nitrate for the Treatment of Dental Sensitivity
Brief Title: Nano-hydroxyapatite With Potassium Nitrate in the Therapy of the Dental Sensitivity
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Università degli Studi di Sassari (Other)
Responsible Party: Principal Investigator, Egle Milia, Prof, Università degli Studi di Sassari
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: DH 2362CE
Record Dates: First submitted 2016-08-04; First posted 2016-09-09 (Estimated); Last update posted 2016-10-26 (Estimated); Status verified 2016-10

CONDITIONS: Dentin Sensitivity
Keywords: nano-hydroxyapatite; potassium nitrate
MeSH Terms: conditions — Dentin Sensitivity | interventions — Sodium Fluoride

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Patients with dentin hypersensitivity (Experimental): Patients with evident clinical signs of dentin hypersensitivity. The following dental materials will be used following the manufacturers' instructions: Cavex Bite&White ExSense and Colgate Protection Caries and Placebo gel.
  In view of the treatment with the desensitizing agents, teeth were randomly assigned into four groups.
  The effectiveness will be evaluated: immediately after application and after 2, 4, 8 weeks.
  Interventions: Other: Cavex Bite&White ExSense; Other: Colgate, Protection Caries; Other: Placebo gel

INTERVENTIONS:
Other: Cavex Bite&White ExSense — a water-based mint aroma gel containing hydroxyapatite and potassium nitrate.
Other: Colgate, Protection Caries — a fluorine-based toothpaste gels
Other: Placebo gel — a glycerin and water gel

SUMMARY:
The chief aim of this study is to evaluate the difference in tooth sensitivity after having used a gel containing nano - hydroxyapatite and potassium nitrate

This randomized double-blind clinical study is designed to compare the efficacy in reducing dentin hypersensitivity of a toothpaste gel containing Nano-hydroxyapatite and potassium nitrate (Cavex Bite & White ExSense, Cavex Holland BV) with a fluoride-based gel toothpaste ( Colgate, Protection Caries, Palmolive SPA ).

Specific objectives :

To evaluate through standardized tests the dental sensitivity before and after the application of toothpastes; To compare the variations of dental sensitivity test and control groups.

Safety:

determination of adverse reactions, such as increased tooth pain and changes in the oral mucosa after application of the materials.

DETAILED DESCRIPTION:
Study Design

The study will be a clinical randomized double-blind trial monocentric.

The sample will be divided into three groups with 35 patients each one.

TREATMENTS NOT ALLOWED

Patients enrolled in the study should not be submitted, for the whole duration of the trial, to local and systemic treatments for dentine hypersensitivity.

Randomization

The randomization process shall be made using a table randomly generated by a computer. The researchers will not be involved in the randomization process.

Data Recording

The study involves the assessment of the following parameters:

During the first visit, data on the overall health and patient's mouth will be collected. All subjects, once included in the study, will receive scaling and polishing treatments.

All these patients will be visited the initial day, once again after 15 days, then after four weeks and eight weeks (end of follow-up). Each subject will be evaluated by the same dentist throughout the course of the trial. During each visit, only the hypersensitive teeth (selected in the beginning of the trial) will be evaluated, so that a minimum of two to a maximum of four sensitive teeth are stimulated by the means of tactile tests and with air spray test.

Tactile test: a sharp dental explorer (EXD 11-12, Hu-Friedy, Chicago, IL, USA) will be dragged on the vestibular side of each tooth, perpendicular to the long axis with a constant force. The test will be repeated three times before recording a score.

Tests air spray: a jet of air will be directed towards the affected tooth area for 1 second from a distance of 10 mm, using a standard air-water syringe, while the adjacent teeth will be isolated with cotton.

The tests with stimuli will be applied in the order previously indicated, with a break of 5 minutes between applications of different stimuli. For tests with stimuli, subjects' responses will be recorded using the following scale:

* 0 - No significant discomfort or awareness of the stimulus;
* 1 - Nuisance, but not acute pain;
* 2 - Acute pain during the application of the stimulus;
* 3 - Acute pain during and after the application of the stimulus.

At each time, a score will be given according to the sensation of pain felt by the patient using a numeric categorical scale with 0-10 parameters (VAS).

Withdrawal of Consent: The patient may at any time withdraw his consent to continue the study. Exit criteria are at the discretion of the researcher: patients who do not show the controls will be excluded from evaluation.

The following dental materials were used following the manufacturers' instructions:

1. Cavex Bite&White ExSense (Cavex Holland BV, RW Haarlem, The Netherlands), a water-based mint aroma gel containing hydroxyapatite and potassium nitrate.
2. Colgate Protection Caries (Palmolive SPA), a fluoride-based gel toothpaste.
3. Placebo gel toothpaste (Baroniestraat, Amsterdam, The Netherlands), a glycerin and water gel.

ELIGIBILITY:
Inclusion Criteria:

* Patients will be considered suitable for the study if they had sensitive teeth showing abrasion, erosion, or recession with the exposure of the cervical dentine.

Exclusion Criteria:

* Teeth with subjective or objective evidence of carious lesions, pulpitis, restorations, premature contact, cracked enamel, active periapical infection, or which had received periodontal surgery or root-planning up to 6 months prior to the investigation will be excluded from the study.
* Professional desensitizing therapy during the previous 3 months, or use of desensitizing toothpaste in the last 6 weeks.
* Patients will be also excluded if they will be under significant medication that could interfere with pain perception (e.g., antidepressants, anti-inflammatory drugs, sedatives, and muscle relaxants).

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2016-03; Primary Completion 2016-05 (Actual); Study Completion 2016-09 (Actual)

PRIMARY OUTCOMES:
Evaluation of change of baseline VAS score at 4 weeks, and 8 Weeks after the treatment | baseline, 4 weeks, and 8 weeks
  The pain experience was assessed by a Visual Analogue Scale (VAS) using the methodology. The VAS scale consisted of a horizontal line that was 100 mm long, on which 'no pain' was marked on the right-hand extremity and 'unbearable pain' on the other. The patients expressed the intensity of the pain experienced by placing a mark at any point along the continuum. The distance, expressed in millimetres, from the right edge of 'no pain' was used as the VAS score. Each patient was asked to rate the perception of discomfort after the application of air via a dental syringe at 45-60 psi, 1 cm at the cervical third of the tooth after removing supragingival plaque with a low- speed handpiece with pumice powder and without fluoride. The adjacent teeth were covered by cotton rolls. The stimulus was delivered until reaction or up to a maximum duration of 10 s by the same examiner with the same equipment yielding similar air pressure each time.

CONTACTS AND LOCATIONS:
Overall Officials: Egle Milia, Prof, Principal Investigator — Università degli Studi di Sassari
Locations (1):
- Complex Operative Unit of Dentistry, Sassari, Sassari, Italy

IPD SHARING:
Plan to Share IPD: No
Not a plan for data sharing has been established. But, for anyone researcher would like to have this information, simply they may request them to us directly.

REFERENCES:
- [Background] Milia E, Castelli G, Bortone A, Sotgiu G, Manunta A, Pinna R, Gallina G. Short-term response of three resin-based materials as desensitizing agents under oral environmental exposure. Acta Odontol Scand. 2013 May-Jul;71(3-4):599-609. doi: 10.3109/00016357.2012.700063. Epub 2012 Aug 15. PMID 22891890
- [Background] Pinna R, Bortone A, Sotgiu G, Dore S, Usai P, Milia E. Clinical evaluation of the efficacy of one self-adhesive composite in dental hypersensitivity. Clin Oral Investig. 2015 Sep;19(7):1663-72. doi: 10.1007/s00784-014-1390-3. Epub 2015 Jan 23. PMID 25609032
- [Background] Vano M, Derchi G, Barone A, Genovesi A, Covani U. Tooth bleaching with hydrogen peroxide and nano-hydroxyapatite: a 9-month follow-up randomized clinical trial. Int J Dent Hyg. 2015 Nov;13(4):301-7. doi: 10.1111/idh.12123. Epub 2015 Jan 20. PMID 25600272
- [Background] Vano M, Derchi G, Barone A, Covani U. Effectiveness of nano-hydroxyapatite toothpaste in reducing dentin hypersensitivity: a double-blind randomized controlled trial. Quintessence Int. 2014 Sep;45(8):703-11. doi: 10.3290/j.qi.a32240. PMID 25019114